CLINICAL TRIAL: NCT00870311
Title: Investigation of Lithium on Signal Transduction, Gene Expression and Brain Myo-Inositol Levels in Manic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Husseini K. Manji, MD, F.R.C.P.C., Wayne State University and National Institute of Mental Health
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H12-48-95; NIMH (MH159107)
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Bipolar Disorder
Keywords: Lithium; Neuroprotection; Neurotrophic; bcl2; gsk3; pkc; MRI; myoinositol; MRS; Alzheimers Disease
MeSH Terms: conditions — Bipolar Disorder; Familial paroxysmal dystonia; Alzheimer Disease | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blinded Lithium (Experimental): Bipolar Disorder patients
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — 300mg PO, three times daily with dose titrated to obtain a therapeutic plasma level of 0.8 to 1.2meq/L) over the first week of treatment. Total duration is a minimum of 3 weeks. Medication is dispensed in the form of blinded research capsules.
  Other Names: Eskalith; Lithonate; Lithane; Lithotabs; Lithobid

SUMMARY:
This study investigates the effects of Lithium treatment on signal transduction pathways, gene expression and brain neurochemistry and structure in patients with Bipolar disorder. It is hypothesized that specific changes in these markers will correlate with lithium treatment responsiveness.

DETAILED DESCRIPTION:
This study investigates the effects of blinded lithium treatment longitudinally in patients with bipolar disorder. At baseline and at multiple time points following the initiation of lithium treatment over 4 or more weeks, measures of signal transduction pathways, gene expression and brain neurochemistry and structure were obtained. It is hypothesized that modulation of these measures will be predictive of lithium treatment responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for Bipolar Mood Disorder determined by DSM-IV (SCID)

Exclusion Criteria:

* Meeting criteria for any other DSM-IV axis I disorder
* Psychoactive substance abuse or dependence within the past 1 year
* Medical conditions placing patients at increased risk for lithium treatment (including renal disease, hepatic disease, hematological disease)
* Devices/implants or conditions which preclude MRI investigation (including cardiac pacemaker/ICD, aneurysm clips, neurostimulator device, metallic fragments in or near the eye,claustrophobia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1996-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Brain myo-inositol levels | 4 weeks

SECONDARY OUTCOMES:
Signal transduction pathway measures | 4 weeks
Gene expression levels | 4 weeks
Brain volume | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Husseini K Manji, MD, Principal Investigator — Wayne State University, National Institute of Mental Health; Debra A Glitz, MD, Principal Investigator — Wayne State University; Gregory J Moore, MD, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University School of Medicine, Detroit, Michigan, United States

REFERENCES:
- [Result] Chen G, Hasanat KA, Bebchuk JM, Moore GJ, Glitz D, Manji HK. Regulation of signal transduction pathways and gene expression by mood stabilizers and antidepressants. Psychosom Med. 1999 Sep-Oct;61(5):599-617. doi: 10.1097/00006842-199909000-00004. PMID 10511011
- [Result] Moore GJ, Bebchuk JM, Parrish JK, Faulk MW, Arfken CL, Strahl-Bevacqua J, Manji HK. Temporal dissociation between lithium-induced changes in frontal lobe myo-inositol and clinical response in manic-depressive illness. Am J Psychiatry. 1999 Dec;156(12):1902-8. doi: 10.1176/ajp.156.12.1902. PMID 10588403
- [Result] Moore GJ, Bebchuk JM, Hasanat K, Chen G, Seraji-Bozorgzad N, Wilds IB, Faulk MW, Koch S, Glitz DA, Jolkovsky L, Manji HK. Lithium increases N-acetyl-aspartate in the human brain: in vivo evidence in support of bcl-2's neurotrophic effects? Biol Psychiatry. 2000 Jul 1;48(1):1-8. doi: 10.1016/s0006-3223(00)00252-3. PMID 10913502
- [Result] Moore GJ, Bebchuk JM, Wilds IB, Chen G, Manji HK. Lithium-induced increase in human brain grey matter. Lancet. 2000 Oct 7;356(9237):1241-2. doi: 10.1016/s0140-6736(00)02793-8. PMID 11072948
- [Derived] Moore GJ, Cortese BM, Glitz DA, Zajac-Benitez C, Quiroz JA, Uhde TW, Drevets WC, Manji HK. A longitudinal study of the effects of lithium treatment on prefrontal and subgenual prefrontal gray matter volume in treatment-responsive bipolar disorder patients. J Clin Psychiatry. 2009 Apr 21;70(5):699-705. doi: 10.4088/JCP.07m03745. PMID 19389332